CLINICAL TRIAL: NCT02924272
Title: An Open-Label, Rollover Protocol for Patients Previously Enrolled in Takeda-Sponsored Ixazomib Studies
Brief Title: Ixazomib Rollover Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Collaborators: Takeda Development Center Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C16027; U1111-1184-2041 (Other: WHO); 2016-001681-28 (EudraCT Number)
Record Dates: First submitted 2016-10-04; First posted 2016-10-05 (Estimated); Results first posted 2025-03-12 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-02

CONDITIONS: Multiple Myeloma; Lymphoma; Amyloidosis
Keywords: Drug Therapy
MeSH Terms: conditions — Multiple Myeloma; Lymphoma; Amyloidosis | interventions — ixazomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ixazomib Monotherapy (Experimental): Participants received ixazomib capsule, orally, at same dose and schedule as they were receiving in the parent study until disease progression, clinical deterioration in the investigator's judgment, experienced an unacceptable toxicity, withdrew consent, pursued an alternative therapy, met other study-specified reasons for discontinuation of study drug, or until the participant was transitioned to ixazomib through commercial channels, including reimbursement for the participant's indication, or up to a maximum of 7 years whichever was sooner.
  Interventions: Drug: Ixazomib
- Ixazomib Combination Therapy (Experimental): Participants received combination therapy with ixazomib capsule, orally and another medication(s) (1 or more of the anticancer agents dexamethasone, lenalidomide or cyclophosphamide) at same dose and schedule as they were receiving in the parent study until disease progression, clinical deterioration in the investigator's judgment, experienced an unacceptable toxicity, withdrew consent, pursued an alternative therapy, met other study-specified reasons for discontinuation of study drug, or until the participant was transitioned to ixazomib through commercial channels, including reimbursement for the participant's indication, or up to a maximum of 6.5 years whichever was sooner.
  Interventions: Drug: Ixazomib

INTERVENTIONS:
Drug: Ixazomib — Ixazomib Capsules
  Other Names: MLN9708; Ninlaro

SUMMARY:
The purpose of this study is to provide continued access to ixazomib and/or other study drugs from an ixazomib parent study.

DETAILED DESCRIPTION:
The drug being tested in this study is called ixazomib. This study will look at the long term safety profile of ixazomib in participants who have previously received and tolerated ixazomib in a Takeda-sponsored clinical study, and in the investigator's opinion and approved by the Takeda medical monitor, may benefit from continued ixazomib therapy.

The study will enroll approximately 250 patients.

All participants will receive ixazomib as a single agent or in combination with other study drugs at same dose and schedule that they were receiving in the parent study until they experience disease progression, clinical deterioration in the investigator's judgment, experience an unacceptable toxicity, withdraw consent, pursue an alternative therapy, meet other study-specified reasons for discontinuation of study drug, or until ixazomib is available to the participant is transitioned to ixazomib/other therapy through commercial channels, including reimbursement for the participant's indication, whichever is sooner.

This multicenter, rollover study will be conducted worldwide. The overall time to participate in this study is up to 7 years. Participants will make multiple visits to the clinic, and a final visit after 30 days of last dose of study drug for a safety assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary written consent must be given before performance of any study-related procedure not part of standard medical care. Participants should consent and enter the study within a maximum of 8 weeks of their last dose of treatment in the parent study or as agreed by the Takeda clinician/designee.
2. Previously treated with ixazomib, background therapy, and/or comparator drugs (including placebo) in a Takeda-sponsored ixazomib parent study. Participants will be eligible to enter the rollover study when:

   1. The parent study is closed or planned to be closed; and
   2. The participant is on ixazomib monotherapy, a combination regimen with ixazomib and other study medication(s), on a placebo combination, or on an alternative arm regimen in a designated ixazomib parent study (i.e., Studies C16003 [NCT00932698], C16005 [NCT01217957], C16006 [NCT01335685], C16007 [NCT01318902], C16008 [NCT01383928], C16010 Global [NCT01564537], C16011 [NCT01659658], C16013 [NCT01645930], C16014 Global [NCT01850524] and Korean Continuation, C16017 [NCT01939899], C16020 [NCT02046070], C16029 [NCT03170882], and C16047 [NCT03439293]); and
   3. In the opinion of the investigator and approved by the Takeda medical monitor, the participant may continue to benefit from treatment with ixazomib and/or another study drug/combination regimen (e.g., response to therapy or stable disease without evidence of disease progression) and has no alternate means to access the study drug(s) (e.g., commercial supply).
3. Agree to continue to practice contraceptive methods as outlined in the parent study.

Exclusion Criteria:

1. The participant meets any of the criteria for treatment discontinuation in the parent study.
2. Female patients who are lactating and breastfeeding or have a positive serum pregnancy test during the eligibility period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2016-12-16 (Actual); Primary Completion 2024-07-03 (Actual); Study Completion 2024-07-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (26):
- United States (4):
  - Emory University, Atlanta, Georgia
  - Appalachian Regional Healthcare, Hazard, Kentucky
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
- UZ Leuven, Leuven, Belgium
- Canada (2):
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - University Health Network, Toronto, Ontario
- China (4):
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - 1st Affiliated Hospital of Zhejiang University, Hangzhou
  - Shanghai Chang Zheng Hospital, Shanghai
- Greece (2):
  - Laiko General Hospital of Athens, Athens, Attica
  - University of Athens Medical School - Regional General Hospital Alexandra, Athens
- Japan (2):
  - Tokyo Metropolitan Komagome Hospital, Bunkyo-Ku, Tokyo
  - Japanese Red Cross Medical Center, Shibuya-Ku, Tokyo
- Poland (4):
  - Samodzielny Publiczny Zaklad Opieki Zdrowotnej Zespol Szpitali Miejskich, Chorzów, Silesian Voivodeship
  - Wojewodzkie Wielospecjalistyczne Centrum Onkologii i Traumatologii im. M. Kopernika w Lodzi, Lodz
  - Centrum Onkologii Ziemi Lubelskiej, Lublin
  - MTZ Clinical Research Sp z o o, Warsaw
- National University Hospital, Singapore, Singapore
- Asan Medical Center - PPDS, Seoul, South Korea
- Spain (2):
  - Hospital Universitario de Donostia, Donostia / San Sebastian
  - Complejo Asistencial Universitario de Salamanca H. Clinico, Salamanca
- Sweden (3):
  - Karolinska Universitetssjukhuset Huddinge, Stockholm, Södermanland County
  - Skanes Universitetssjukhus Lund, Lund
  - Karolinska Universitetssjukhuset Solna, Stockholm

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at various investigative sites globally from 16 December 2016 to 03 July 2024.
Pre-assignment Details: Participants who had previously received and tolerated treatment in ixazomib parent studies (C16003 [NCT00932698], C16005 [NCT01217957], C16006 [NCT01335685],C16007 [NCT01318902],C16008 [NCT01383928],C16010 Global [NCT01564537],C16011 [NCT01659658],C16013 [NCT01645930],C16014 Global [NCT01850524] and Korean Continuation,C16017 [NCT01939899],C16020 [NCT02046070],C16029 [NCT03170882], or C16047 [NCT03439293]), and in investigator's opinion could benefit from continued therapy were enrolled.
Groups:
- Ixazomib Monotherapy: Participants received ixazomib capsule, orally, at same dose and schedule as they were receiving in the parent study until disease progression, clinical deterioration in the investigator's judgment, experienced an unacceptable toxicity, withdrew consent, pursued an alternative therapy, meet other study-specified reasons for discontinuation of study drug, or until the participant was transitioned to ixazomib through commercial channels, including reimbursement for the participant's indication, or up to a maximum of 7 years whichever was sooner.
Period: Overall Study
Arm/Group | Ixazomib Monotherapy | Ixazomib Combination Therapy
Started | 23 | 9
Completed | 0 | 0
Not Completed | 23 | 9
Not completed — Site Terminated by Sponsor | 4 | 1
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Adverse Event | 3 | 0
Not completed — Progressive Disease | 11 | 8
Not completed — Clinical Deterioration | 1 | 0
Not completed — Death | 1 | 0
Not completed — Reason Not Specified | 1 | 0

BASELINE CHARACTERISTICS:
Population: The Safety Population included all enrolled participants who received at least 1 dose of ixazomib.
Groups:
- Total: Total of all reporting groups
Arm/Group | Ixazomib Monotherapy | Ixazomib Combination Therapy | Total
Number analyzed (Participants) | 23 | 9 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 75.1 (6.45) | 64.6 (9.53) | 72.2 (8.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 5 | 16
  Male | 12 | 4 | 16
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs)
Description: An adverse event (AE) is defined as any untoward medical occurrence in a participant administered a pharmaceutical product; the untoward medical occurrence does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product whether or not it is related to the medicinal product. An SAE is any untoward medical occurrence that at any dose: a) results in death; b) is life-threatening (refers to an AE in which the participant was at risk of death at the time of the event. It does not refer to an event which hypothetically might have caused death if it were more severe); c) requires inpatient hospitalization or prolongation of an existing hospitalization; d) results in persistent or significant disability or incapacity; e) is a congenital anomaly/birth defect; f) is a medically important event.
Time Frame: Up to 7 years
Population: Safety Population included all enrolled participants who received at least 1 dose of ixazomib.
Measure: Count of Participants; unit: Participants
Arm/Group | Ixazomib Monotherapy | Ixazomib Combination Therapy
Number analyzed (Participants) | 23 | 9
Participants | 12 | 4

2. Primary Outcome: Number of Participants With ≥ Grade 3 AEs
Description: An AE is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (e.g., a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, whether or not it is considered related to the drug. The severity grade was evaluated as per the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5.0. Grade 3: severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care activities of daily living (ADL), Grade 4: life-threatening consequences; urgent intervention indicated. Grade 5 was: death related to AE.
Time Frame: Up to 7 years
Population: Safety Population included all enrolled participants who received at least 1 dose of ixazomib.
Measure: Count of Participants; unit: Participants
Arm/Group | Ixazomib Monotherapy | Ixazomib Combination Therapy
Number analyzed (Participants) | 23 | 9
Participants | 13 | 5

3. Primary Outcome: Number of Participants With ≥ Grade 2 Peripheral Neuropathy
Description: Severity grade was evaluated based on CTCAE version 5.0. Grade 2: moderate symptoms; limiting instrumental activities of daily living. Grade 3: severe or medically significant; limiting self-care activities of daily living. Grade 4: life threatening consequences; urgent intervention indicated.
Time Frame: Up to 7 years
Population: Safety Population included all enrolled participants who received at least 1 dose of ixazomib.
Measure: Count of Participants; unit: Participants
Arm/Group | Ixazomib Monotherapy | Ixazomib Combination Therapy
Number analyzed (Participants) | 23 | 9
Participants | 2 | 0

4. Primary Outcome: Number of Participants With New Primary Malignancies
Time Frame: Up to 7 years
Population: Safety Population included all enrolled participants who received at least 1 dose of ixazomib.
Measure: Count of Participants; unit: Participants
Arm/Group | Ixazomib Monotherapy | Ixazomib Combination Therapy
Number analyzed (Participants) | 23 | 9
Participants | 3 | 1

5. Primary Outcome: Number of Participants With Any AE Resulting in Dose Modification or Discontinuation of Any Study Drug
Description: An AE means any untoward medical occurrence in a participant administered a pharmaceutical product; the untoward medical occurrence does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product whether or not it is related to the medicinal product.
Time Frame: Up to 7 years
Population: Safety Population included all enrolled participants who received at least 1 dose of ixazomib.
Measure: Count of Participants; unit: Participants
Arm/Group | Ixazomib Monotherapy | Ixazomib Combination Therapy
Number analyzed (Participants) | 23 | 9
Participants
  AE Resulting in Dose Modification | 12 | 7
  AE Resulting in Discontinuation of Study Drug | 4 | 1

6. Primary Outcome: Number of Participants With Any Other AE That in the Opinion of the Investigator is a Clinically Significant Event
Description: An AE means any untoward medical occurrence in a participant administered a pharmaceutical product; the untoward medical occurrence does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product whether or not it is related to the medicinal product. Any AE interpreted by the investigator as a clinically significant event was reported.
Time Frame: Up to 7 years
Population: Safety Population included all enrolled participants who received at least 1 dose of ixazomib.
Measure: Count of Participants; unit: Participants
Arm/Group | Ixazomib Monotherapy | Ixazomib Combination Therapy
Number analyzed (Participants) | 23 | 9
Participants | 15 | 7

ADVERSE EVENTS:
Time Frame: Up to 7 years
Description: The Safety Population included all enrolled participants who received at least 1 dose of ixazomib.
Arm/Group | Ixazomib Monotherapy | Ixazomib Combination Therapy
All-Cause Mortality (participants affected / at risk) | 1/23 | 0/9
Serious Adverse Events (participants affected / at risk) | 12/23 | 4/9
Other Adverse Events (participants affected / at risk) | 9/23 | 6/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ixazomib Monotherapy (N=23) | Ixazomib Combination Therapy (N=9)
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Angina unstable (Cardiac disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Balance disorder (Nervous system disorders) | 1 | 0
Bladder injury (Injury, poisoning and procedural complications) | 1 | 0
Bronchiolitis (Infections and infestations) | 1 | 0
COVID-19 pneumonia (Infections and infestations) | 0 | 1
Cardiac failure (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Osteomyelitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 2 | 3
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0
Sebaceous carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Tuberculous pleurisy (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ixazomib Monotherapy (N=23) | Ixazomib Combination Therapy (N=9)
Alanine aminotransferase increased (Investigations) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 3
Ankle fracture (Injury, poisoning and procedural complications) | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 2
COVID-19 (Infections and infestations) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 1
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 1
Hepatotoxicity (Hepatobiliary disorders) | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 1
Hypertension (Vascular disorders) | 4 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0
Pneumonia (Infections and infestations) | 1 | 1
Tooth abscess (Infections and infestations) | 0 | 1
Tooth infection (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 3 | 3
Vomiting (Gastrointestinal disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-06-03): https://cdn.clinicaltrials.gov/large-docs/72/NCT02924272/Prot_000.pdf
  • Statistical Analysis Plan (2023-09-15): https://cdn.clinicaltrials.gov/large-docs/72/NCT02924272/SAP_001.pdf